CLINICAL TRIAL: NCT03624491
Title: Mechanical Ventilation Guided By Transpulmonary and Airway Driving Pressures in the Setting of Intra-abdominal Hypertension
Brief Title: Esophageal Balloon Measurements to Better Characterize Thoraco-abdominal Interrelationship Mechanics.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Richard A. Oeckler, M.D., Ph.D., Assistant Professor of Medicine and Physiology-Critical Care, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-007482
Record Dates: First submitted 2017-11-02; First posted 2018-08-10 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Surgery

STUDY DESIGN:
Intervention Model Description: Randomization to two different groups.
Masking Description: This is a prospective, open label, randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care mechanical ventilation (No Intervention): Anesthesia and surgical procedures will be performed following standard of care for mechanical ventilation during surgery.
- Transpulmonary pressure guided mechanical ventilation (Active Comparator): Same treatment as the control group with the addition of esophageal pressure measurements used to guide mechanical ventilation during surgery.
  Interventions: Other: Esophageal pressure measurement guided ventilation

INTERVENTIONS:
Other: Esophageal pressure measurement guided ventilation — Use of esophageal pressure measurements to guide mechanical ventilation
  Arms: Transpulmonary pressure guided mechanical ventilation

SUMMARY:
Esophageal pressure measurements in surgical patients requiring mechanical ventilation during abdominal laparoscopic or robotic surgeries requiring intra-abdominal insufflation.

DETAILED DESCRIPTION:
Decades of research and clinical observation in mechanical ventilation have demonstrated unequivocally that tidal volume (VT), plateau pressure (PPLAT) and PEEP (positive end-expiratory pressure) influence ventilator induced lung injury. Clinicians, however, have struggled in the attempt to find a single indicator of safety and risk. Recent analyses of the large multi-center randomized trials database suggest that Airway Driving Pressure (ADP) and Trans pulmonary Driving Pressure (DTP) are the variables of greatest importance and therefore the best single parameters on which to focus. In attempting to define their optimal values and their correlation between each other in the setting of intra-abdominal hypertension, we would like to compare standard of care mechanical ventilation (control) with mechanical ventilation guided by DTP and ADP (intervention) in patients undergoing abdominal laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring mechanical ventilation for abdominal laparoscopic and robotic surgeries.
* Patients who are passively ventilated (no respiratory efforts) as a result of the sedation plan determined entirely by the primary anesthesia team --research team will not influence or participate on the sedation protocol plan or implementation.
* Patients who are clinically stable and able to tolerate the changes in position that are routinely conducted as part of the standard of care in the operative room.
* Patient/responsible family member signing the informed consent must speak English.

Exclusion criteria:

* Patients with open abdomen prior to surgical procedures.
* Females of childbearing age (18-50) with the potential to become pregnant and no clinically documented negative pregnancy test.
* Patients with clinically evident spontaneous breathing efforts (ventilator wave forms) during surgical procedure.
* Patients with clinical suspicion of elevated intra-cranial pressure (requiring head elevation).
* Contraindication to body position change, as dictated by surgery-specific protocol.
* Unstable cardio-respiratory insufficiency.
* Age less than 18 years.
* Cuff leak in endotracheal / tracheostomy tube.
* Patient/responsible family member unable to understand the informed consent in English.
* Patient with contraindication for nasogastric tube placement:

  * Severe midface trauma
  * Recent nasopharyngeal surgery
  * Coagulation abnormality
  * Esophageal varices, stricture, ulcerations, or tumors
  * Recent banding of esophageal varices
  * Alkaline ingestion
  * Diverticulitis,
  * Sinusitis, epistaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Airway driving pressure guided mechanical ventilation determined by esophageal balloon catheter measurements. | Through study completion, an average of one year
  Optimizing the relationship between intra-abdominal pressure and both airway driving pressure and trans pulmonary driving pressure utilizing esophageal balloon measurements to guide mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Oeckler, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayoclinic.org/